CLINICAL TRIAL: NCT04929145
Title: Microbiome Benchmarking to Identify Perturbations in Multiple Sclerosis I
Brief Title: The Gut Microbiome in Adult Multiple Sclerosis
Acronym: MICROMS5Y
Status: Completed | Type: Observational
Sponsor: National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Marie D'hooghe, Neurologist/Clinical Professor, National MS Center Melsbroek
Other Study IDs: MICROMS5Y
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: gut microbiome
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal specimens from patients will be collected with standard kits and frozen for analysis.
  A blood sample of 10 ml will be drawn from a peripheral vein for the analysis of IL-1beta and Il-17 (proinflammatory cytokines) and and IL-10 (anti-inflammatory cytokine), and a range of amino acids (released by the gut) through HPLC. A serum sample will be deep frozen for further analyses.
  Some hair will be cut at the vertex posterior, close to the skull. A number of 5-10 hairs, corresponding to 5 mg, will be collected and stored in a cool place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MICROMS: No intervention will be administered. Stool, hair, and blood samples will be collected at baseline and three months post baseline. Clinical follow-up will occur at year 1, 2, and 4.5 (neurological consultation) and in-between visits (regular follow-up).

SUMMARY:
This study aims to assess the following research questions:

1. Map and benchmark the gut microbiome of patients with RRMS, and PPMS versus matched healthy controls
2. Determine whether RRMS or PPMS have a unique bias for a gut microbiome classification recently characterized.
3. Search for relationship with inflammation, amino acid plasma levels, heart rate variability (vagus nerve tone) and hair cortisol as a biological marker of chronic stress
4. Determine whether the gut microbiome is different in MS patients during a relapse.
5. Determine whether the gut microbiome remains stable after 3 months

DETAILED DESCRIPTION:
This study is a prospective multi-center cohort study (University Hospital Brussels, National Multiple Sclerosis Center Melsbroek). This is an exploratory study and there is no specific outcome on which a power calculation can be made. We will include different subgroups of patients with MS: stable non-benign RRMS, PPMS, benign MS [Benign MS is defined as RRMS with an EDSS ≤ 3, 15 years after disease onset], RRMS during a relapse (before the administration of corticosteroids) [Relapses are defined as the development of new or recurrent neurologic symptoms not associated with fever or infection or change in medication, lasting at least 24 hours, and accompanied by new, objective neurologic findings]. Age and sex matched healthy controls will be included as well. All participants will provide a faecal, hair, and blood sample twice (baseline and after 3 months). Patients will be assessed clinically at baseline, 3 months after baseline, and approximately 1, 2, 4.5 years after baseline.

The results of this study have the potential to identify novel simple strategies to strengthen or alter the microbiome ecosystem and strengthen the overall treatment process. In case of a positive result, this would form the basis for a follow-up study on medical modulation of the microbiome with the aim of finding new treatment options for MS.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. RRMS or PPMS, as defined by the McDonald criteria.
3. Ages 18-65 years.
4. EDSS < 7
5. Treatment with IFN-beta

Exclusion Criteria:

1. SPMS without relapses during the past year at screening.
2. Use of high dose systemic steroids within the last 2 months.
3. Gastrointestinal disease, such as inflammatory bowel disease
4. Use of antibiotics within the last 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an exploratory study and there is no specific outcome on which a power calculation can be made. We included 122 patients with MS and 30 age and sex matched healthy controls as well.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Sustained disability worsening | 5 years
  Sustained disability worsening will be assessed using the Expanded Disability Status Scale (EDSS)-Plus outcome. This is a composite measure that assesses disability worsening based on changes of the EDSS score (difference of at least 1.5;1.0;0.5 depending on baseline score), the timed 25-foot walk (T25FW) score (>=20%), and the 9-hole peg test (9-HPT) score (>=20%). If worsening of any of these measures occurred, the patient has clinically deteriorated according to the EDSS-Plus outcome.

SECONDARY OUTCOMES:
Clinical evidence for active disease | 5 years
  Time to first relapse (after baseline) will be reported for all patients. Annualized relapse frequency

CONTACTS AND LOCATIONS:
Overall Officials: Marie D'hooghe, M.D., Principal Investigator — National MS Center Melsbroek
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussel-Hoofdstedelijk-Gewest
  - Nationaal Multiple Sclerose Centrum Melsbroek, Melsbroek, Vlaams-Brabant

REFERENCES:
- [Derived] Devolder L, Pauwels A, Van Remoortel A, Falony G, Vieira-Silva S, Nagels G, De Keyser J, Raes J, D'Hooghe MB. Gut microbiome composition is associated with long-term disability worsening in multiple sclerosis. Gut Microbes. 2023 Jan-Dec;15(1):2180316. doi: 10.1080/19490976.2023.2180316. PMID 36803643